CLINICAL TRIAL: NCT04677673
Title: Neoadjuvant Chemotherapy Plus Surgery Versus Surgery First For Elderly Gastric Cancer Patients
Acronym: RJGC-Senile
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BIRENDRA KUMAR SAH (Other)
Responsible Party: Sponsor-Investigator, BIRENDRA KUMAR SAH, Principal Investigator, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dragon Senile
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Gastric Cancer; Chemotherapy Effect; Elderly Patients; Surgery
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC PLUS SURGERY (Experimental): Patients receive three cycles of the modified dose of TGO plus oxaliplatin before curative gastrectomy.
  Interventions: Drug: Chemotherapy
- SURGERY FIRST (Active Comparator): Patients undergo curative gastrectomy without any prior chemotherapy.
  Interventions: Procedure: Curative gastrectomy

INTERVENTIONS:
Drug: Chemotherapy — Modified SOX Chemotherapy regimen A cycle consists of Day 1: Oxaliplatin 100mg/M2 intravenous Day 1-14 Tegafur gimeracil oteracil potassium capsule 60mg/M2 oral (twice daily) Repeated every 22nd day
  Other Names: Modified SOX
  Arms: NAC PLUS SURGERY
Procedure: Curative gastrectomy — Radical gastrectomy with D2 lymph node dissection
  Arms: SURGERY FIRST

SUMMARY:
The main purpose of this study is to compare the feasibility and efficacy of neoadjuvant chemotherapy (modified SOX) for elderly patients with locally advanced gastric cancer.

DETAILED DESCRIPTION:
DRAGON SENILE research, Neoadjuvant Chemotherapy plus Surgery versus surgery first for elderly Gastric Cancer patients, is an investigator-initiated; phase II/III, open-label, randomized controlled study. The main purpose of this study is to compare the feasibility and efficacy of neoadjuvant chemotherapy (modified SOX) for elderly patients with locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histology confirmed non-obstructive adenocarcinoma of the stomach or esophagogastric junction.
* Clinical stage: cTNM: stage III
* Performance status: Eastern Cooperative Oncology Group ECOG ≤ 2 (normal to symptomatic but in bed less than half the day)
* Clinically fit for systemic chemotherapy and gastric cancer surgery, i.e. adequate renal, hepatic, hematologic, and pulmonary function.
* Written informed consent

Exclusion Criteria:

* Clinically unfit for systemic chemotherapy and gastric cancer surgery, i.e. uncontrolled cardiac disease, or other clinically significant uncontrolled comorbidities, unable to undergo general anesthesia
* Distant metastases (including retroperitoneal lymph node)
* Locally advanced inoperable disease (Clinical assessment)
* Relapse of gastric cancer
* Malignant secondary disease
* Prior chemo or radiotherapy
* Inclusion in another clinical trial
* Known contraindications or hypersensitivity for planned chemotherapy

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Five years
  Time from randomization to death from any cause

SECONDARY OUTCOMES:
Completion rate of planned NAC | Three months
  Completion rate of planned chemotherapy before surgery.
Percentage of Grade 3/4 hematological adverse events | Three months
  Percentage of Grade 3/4 hematological adverse events during neoadjuvant chemotherapy
Pathological response | Four months
  Total percentage of patients with pathological complete tumor regression (TRG1a) and sub-total tumor regression (TRG1b) in the primary tumor
Disease-free survival (DFS) | Two years
  Time from randomization to relapse of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Zhenggang Zhu, Study Chair — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No